CLINICAL TRIAL: NCT06403774
Title: Effect of Two Different Bowel Preparation Methods on Outcomes After Hemorrhoidectomy
Brief Title: Bowel Preparation Before Hemorrhoidectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Bediye Öztaş, Principal investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 913715751
Record Dates: First submitted 2024-04-20; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: HEMORRHOIDECTOMY
Keywords: HEMORRHOIDECTOMY; BOWEL PREPARATION; PAIN; COMFORT
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: TWO DIFFERENT BOWEL PREPARATION METHODS WILL BE COMPARED IN PATIENTS WHO WILL HAVE HEMORRHOIDECTOMY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group that will undergo bowel preparation using laxatives (Two bowel X-M Solution 250 ml.) (Experimental): Bowel preparation will be made using a laxative (Two bowel X-M Solution 250 ml.)
  Interventions: Drug: Group that will undergo bowel preparation using laxatives (Two bowel X-M Solution 250 ml.)
- Group that will undergo bowel preparation using enema (Two bowel E.S. Enema ) (Experimental): Bowel preparation will be made using enema (Two bowel E.S. Enema )
  Interventions: Drug: Group that will undergo bowel preparation using enema (Two bowel E.S. Enema )

INTERVENTIONS:
Drug: Group that will undergo bowel preparation using laxatives (Two bowel X-M Solution 250 ml.) — A laxatives (Two bowel X-M Solution 250 ml.) will be applied for bowel preparation before hemorrhoidectomy. The drug was given to the patient at 3 o'clock (p.m.)before the surgery by mixing it with 1500ml of water.
  Arms: Group that will undergo bowel preparation using laxatives (Two bowel X-M Solution 250 ml.)
Drug: Group that will undergo bowel preparation using enema (Two bowel E.S. Enema ) — An enema (Two bowel E.S. Enema ) will be applied for bowel preparation before hemorrhoidectomy.The drug was administered to the patient at 00 o'clock (a.m.) and 06 o'clock (a.m.) before the surgery.
  Arms: Group that will undergo bowel preparation using enema (Two bowel E.S. Enema )

SUMMARY:
The purpose of this research; To evaluate the effect of preoperative bowel preparation on post-hemorrhoidectomy outcomes. Bowel preparation is a routine practice before surgery in anorectal diseases. This study aims to evaluate the effect of bowel preparation using laxatives or enemas on the patient postoperative pain, analgesic consumption amount, comfort, first defecation time and satisfaction, and to evaluate the satisfaction of the surgical team.

DETAILED DESCRIPTION:
The study is planned as a semi-experimental. The effect of bowel preparation using laxatives or enemas on postoperative pain, analgesic consumption, comfort and satisfaction will be evaluated. Criteria for inclusion in the research; Being a patient who will undergo hemorrhoidectomy with spinal anesthesia and agreeing to participate in the study are the exclusion criteria; Refusal to participate in the research was determined as. Following the admission of the patient, who is planned to undergo hemorrhoidectomy, to the clinic, the patient will be interviewed, the purpose of the study will be explained and he/she will be invited to participate in the study. Written consent will be obtained from patients who agree to participate in the research.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient who will undergo hemorrhoidectomy surgery with spinal anesthesia
* Agreeing to participate in the study

Exclusion Criteria:

* Not accepting participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain level | postoperative 2, 6, 10, 20, 24. hours and at the first defecation assessed up to 72 hours
  To evaluate pain; A numerical rating scale will be used, numbered 0-10, 0: no pain, 10: unbearable pain (1-3 mild, 4-6 moderate, 7-10 severe).

SECONDARY OUTCOMES:
Analgesic consumption amount | First 24 hours postoperatively
  Total amount of analgesic used in the first 24 hours postoperatively
Comfort level | It will be evaluated once at the 24th postoperative hour.
  To evaluate comfort; Perianesthesia comfort scale will be used.Perianesthesia Comfort Scale (PCS) consists of 24 items that reflect the individual's general thought process about the perianesthesia period and question his/her self-conception and feelings.
  Each statement in the scale has a Likert-type scoring ranging from 1-6, from "strongly disagree" to "strongly agree".
  The highest total score that can be obtained from the scale is 144, and the lowest total score is 24.
  The average value is determined by dividing the total score obtained by the number of scale items and the result is stated in the 1-6 distribution.
  A low score indicates poor comfort and a high score indicates good comfort.
Satisfaction level of patients | It will be evaluated once at the 24th postoperative hour.
  To evaluate the satisfaction of patients and the surgical team; A numerical evaluation scale (numbered between 0-10, 0: not at all satisfied, 10: very satisfied) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: bediye oztas, phd, Principal Investigator — nursing
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing will be possible when the work is published.

REFERENCES:
- [Background] • De la Garza M.,.Counihan T.C. Complications of hemorrhoid surgery. Seminars in Colon and Rectal Surgery 24 (2013) 96-102
- [Background] Sammour T, Barazanchi AW, Hill AG; PROSPECT group (Collaborators). Evidence-Based Management of Pain After Excisional Haemorrhoidectomy Surgery: A PROSPECT Review Update. World J Surg. 2017 Feb;41(2):603-614. doi: 10.1007/s00268-016-3737-1. PMID 27766395